CLINICAL TRIAL: NCT05427435
Title: Prospective Single-centre Study to Evaluate the Feasibility of Ethanolization of Vein of Marshall With a Specific Catheter in the Ablation of Atrial Fibrillation
Brief Title: Feasibility of Ethanolization of Vein of Marshall With Specific Catheter in Atrial Fibrillation Ablation
Acronym: Innov Marshall
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2021/18
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
Keywords: Persistent atrial fibrillation; Pulmonary vein isolation; Catheter ablation; Ethanolization; Ligament of Marshall; Vein of Marshall
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: prospective single arm monocentric evaluation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Marshall ethanolisation with specific catheter (Experimental): Patients will undergo the destruction of Marshall bundles by ethanol infusion with the specific catheter
  Interventions: Device: Marshall ethanolisation

INTERVENTIONS:
Device: Marshall ethanolisation — Destruction of Marshall bundles by ethanol 96% infusion (3 separate injections of 3.3ml)

SUMMARY:
In patients with persistent AF (PsAF), ablation limited to pulmonary vein (PV) isolation is the most straightforward approach, but results only in 50% of arrhythmia freedom at 1 year follow-up. Substrate modification strategies have failed to demonstrate their superiority with variable reported success rate. The Marshall network is a highly arrhythmogenic structure that has not been systematically targeted so far, probably because of the absence of dedicated tools to make its ablation simple and easy. We sought to investigate the use of a specific catheter for visualization and ethanolization of vein of Marshall allowing to systematically include this target in the ablation set.

The main objective of this study is to demonstrate the feasibility to use the Targeted Endovascular Delivery (TED) catheter specifically for visualization and ethanolization of vein of Marshall.

ELIGIBILITY:
Inclusion Criteria:

* Suitable candidate for catheter ablation of atrial fibrillation defined as:

  * history of symptomatic persistent atrial fibrillation
  * Redo procedure for persistent AF or paroxysmal AF with isolated PV and no history of ethanol infusion in the VOM.
* Age > 18 years of both genders
* Patient affiliated or beneficiary of social security scheme
* Free, informed and written consent signed by the participant and the principal investigator (at least at the inclusion date and before all exams required for the clinical research)
* Effective contraception for women of childbearing potential

Exclusion Criteria:

* Minor
* Documented left atrial thrombus or another abnormality which precludes catheter introduction
* Contraindication to anticoagulation therapy (heparin, warfarin, or novel oral anticoagulant [NOAC]
* Contraindication to iodinated contrast product XENETIX® (iobitridol hypersensivity or at one of these excipients, history of major immediate reaction or cutaneous reaction to XENETIX® infusion, thyrotoxicosis)
* Hypersensitivity to ethanol
* Unstable angina or ongoing myocardial ischemia
* Myocardial infarction within 3 months prior to inclusion
* Congenital heart disease, where the underlying abnormality increases the ablation risk
* Severe bleeding, clotting or thrombotic disorder
* Pregnant, parturient or nursing women
* Unable or unwilling to provide written informed consent
* Patient detained by judicial or administrative order
* Patient under psychiatric care
* Patient admitted in a social or healthcare establishment for any purpose other than the research
* Subject to a legal protection order (guardianship, patient under legal protection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2027-05-16 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Acute success rate of the procedure | 12 months
  Success rate complete realization of ethanolization procedure

SECONDARY OUTCOMES:
Total duration of ethanolization procedure | 12 months
  Time between the entry and the removal of the catheter
Time to visualization of Vein of Marshall | 12 months
  Time between 1st injection of iodine (contrast media) and time of visualization of Vein of Marshall
Duration of balloon positioning | 12 months
  Time from the 1st injection of iodine to the 1st injection of ethanol
Total X Ray duration and radiation dose | 12 months
  Time of exposure to X Ray and total of received radiation dose
Incidence of Vein of Marshall dissection | 12 months
  Rate of Vein of Marshall dissection
Incidence of periprocedural complications related to ethanolization | 12 months
  Number and rate of adverse events related to ethanolization
Incidence of complications related to catheter | 12 months
  Number and rate of adverse events related to the catheter or its procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MD DERVAL, Principal Investigator — Study Principal Investigator
Locations (1):
- CHU de Bordeaux, Pessac, France